CLINICAL TRIAL: NCT02372331
Title: The Effect of ERAS (Enhanced Recovery After Surgery) on Pancreaticoduodenectomy
Brief Title: The Effect of ERAS on Pancreaticoduodenectomy
Acronym: ERAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Dae Wook Hwang, Assistant professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERAS
Record Dates: First submitted 2015-02-12; First posted 2015-02-26 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Periampullary Tumor
Keywords: pancreaticoduodenectomy; ERAS; Whipple's operation; Fast track

STUDY DESIGN:
Intervention Model Description: Two study groups (Control (conventional) group and study (intervention) group) were randomly allocated and assigned to one of two groups in parallel for the whole duration of this study.
Who Masked: Outcomes Assessor
Masking Description: The evaluation and judgement for morbidity (primary endpoint) / mortality (secondary endpoint) was made by Morbidity and Mortality Committee in our division. Committee members were blinded about knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional perioperative management (No Intervention): * Preop usual biliary drainage
  * Preop smoking and alcohol
  * Preop parenteral nutrition
  * Oral bowel preparation (mechanical bowel preparation )
  * Preoperative fasting > 12 hours
  * Pre-anesthetic medication
  * Anti-thrombotic prophylaxis
  * Antimicrobial prophylaxis and skin preparation
  * Intravenous analgesia : PCA
  * Prevention of postoperative nausea and vomiting (PONV) (X)
  * Incision : surgeon direction
  * Avoiding hypothermia
  * Nasogastric intubation (O)
  * Postop glycemic control
  * Positive fluid balance
  * Perianastomotic drain removal over POD #5
  * Somatostatin analogues
  * Transurethral catheter removal
  * Delayed gastric emptying(DGE) (+) , parenteral nutrition (+)
  * Postop routine artificial nutrition (O), soft diet at POD #5
  * Early and scheduled mobilization
- ERAS perioperative management (Experimental): * behavioral intervention (counselling, audit)
  * dietary supplement
  * procedure (preoperative and postoperative)
  * drug
  Interventions: Other: ERAS perioperative management

INTERVENTIONS:
Other: ERAS perioperative management — * Preop Counseling
  * Preop biliary drainage (X) when Serum Total bilirubin < 14.62mg/dl and cholangitis (-)
  * Preop enteral nutrition
  * Oral bowel preparation (mechanical bowel preparation ) (X)
  * Preop fasting < 6 hours
  * Prevention of postoperative nausea and vomiting (PONV) (O)
  * Nasogastric intubation (X)
  * Near-zero fluid balance
  * Somatostatin analogues (X)
  * Postop routine artificial nutrition (X), soft diet at POD #2
  * Audit
  * Other items are same as conventional
  Other Names: Fast tract
  Arms: ERAS perioperative management

SUMMARY:
Enhanced Recovery After Surgery (ERAS) is not the program that aim to reduce postoperative hospital stay, but the multimodal strategies that aim to attenuate the loss of, and improve the restoration of,functional capacity after surgery on evidence-based medicine. The benefits of ERAS is proved in many surgical procedures, such as upper gastrointestinal surgery and colorectal surgery. However, pancreaticoduodenectomy (PD, Whipple's operation) is still one of most complex abdominal surgery, and there is no evidence that ERAS is beneficial on PD.

This study investigate the clinical effectiveness of ERAS on PD.

DETAILED DESCRIPTION:
* This study conduct totally 276 patients who underwent PD with borderline or malignant periampullary tumor. The patients divided into two groups. One group take conventional, experienced-based perioperative management, the other group take perioperative management based on ERAS protocol. Applied ERAS protocol is based on "Guidelines for Perioperative Care for Pancreaticoduodenectomy: Ehanced Recovery After Surgery Society Recommendations.
* The outcomes are analyzed for short-term surgical outcomes including operative factors, nutritional status, morbidity, mortality, length of stay, readmission, etc.
* Among all subjects who were randomized and started any study intervention (ERAS or standard perioperative management), the patients who underwent pancreaticoduodenectomy were included as the Full analysis set (FAS). All subjects who didn't undergo pancreaticoduodenectomy were excluded from this study.
* Besides, as all subjects who were randomized and received any study intervention were obliged to follow the study protocol and monitored for best compliance, per-protocol set or safety set were not defined differently

ELIGIBILITY:
Inclusion Criteria:

* >18 years old or <75 years old
* ECOG 0-2
* resectable periampullary cancer or borderline malignancy
* no distant metastasis
* no functional disturbance in bone marrow; WBC at least 3,000/mm3 or absolute neutrophil count at least 1,500/mm3, Platelet count at least 125,000/mm3
* no functional disturtance in liver; Bilirubin less than 2.5 mg/dL AST less than 5 times upper limit of normal
* no function disturbance in kidney; Creatinine no greater than 1.5 times upper limit of normal
* informed consent

Exclusion Criteria:

* distant metastasis (+) or recurred periampullary tumor
* active or uncontrolled infection
* uncontrolled psychiatric or neurologic problems
* alcohol or other drug addiction
* already enrolled patient in other study which affect this study
* the patient who is impossible to allow investigator's order
* pregnant or the possibility of pregnancy (+)
* uncontrolled cardiopulmonary disease
* moderate to severe comorbidity which affect on the quality of life and nutritional status (liver cirrhosis, end stage renal disease, heart failure, etc.)
* previous history of major gastrointestinal surgery (gastrectomy, colectomy, etc.)
* in preoperative period, expected combined resection of other gastrointestinal organ including portal vein

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2015-03-04 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-26 (Actual)

PRIMARY OUTCOMES:
Morbidity | 3 months
  The incidence of operation-related morbidity

SECONDARY OUTCOMES:
Mortality | 3 months
  The incidence of 30 days mortality and in-hospital mortality
length of stay | 3 months
  postoperative length of stay
nutritional status | 3 months
  The nutritional status would be analyzed by the comparison of PG-SGA score, body mass index and assessment of daily oral intake at preoperative, before discharge and postoperative 2~3months.

CONTACTS AND LOCATIONS:
Overall Officials: Dae Wook Hwang, M.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
At initial status of this study, IRB was approved at limited data access only.

REFERENCES:
- [Background] American Society of Anesthesiologists Committee. Practice guidelines for preoperative fasting and the use of pharmacologic agents to reduce the risk of pulmonary aspiration: application to healthy patients undergoing elective procedures: an updated report by the American Society of Anesthesiologists Committee on Standards and Practice Parameters. Anesthesiology. 2011 Mar;114(3):495-511. doi: 10.1097/ALN.0b013e3181fcbfd9. No abstract available. PMID 21307770
- [Background] Balzano G, Zerbi A, Braga M, Rocchetti S, Beneduce AA, Di Carlo V. Fast-track recovery programme after pancreatico- duodenectomy reduces delayed gastric emptying. Br J Surg. 2008 Nov;95(11):1387-93. doi: 10.1002/bjs.6324. PMID 18844251
- [Background] Berberat PO, Ingold H, Gulbinas A, Kleeff J, Muller MW, Gutt C, Weigand M, Friess H, Buchler MW. Fast track--different implications in pancreatic surgery. J Gastrointest Surg. 2007 Jul;11(7):880-7. doi: 10.1007/s11605-007-0167-2. PMID 17440787
- [Background] di Sebastiano P, Festa L, De Bonis A, Ciuffreda A, Valvano MR, Andriulli A, di Mola FF. A modified fast-track program for pancreatic surgery: a prospective single-center experience. Langenbecks Arch Surg. 2011 Mar;396(3):345-51. doi: 10.1007/s00423-010-0707-1. Epub 2010 Aug 12. PMID 20703500
- [Background] Fearon KC, Ljungqvist O, Von Meyenfeldt M, Revhaug A, Dejong CH, Lassen K, Nygren J, Hausel J, Soop M, Andersen J, Kehlet H. Enhanced recovery after surgery: a consensus review of clinical care for patients undergoing colonic resection. Clin Nutr. 2005 Jun;24(3):466-77. doi: 10.1016/j.clnu.2005.02.002. Epub 2005 Apr 21. PMID 15896435
- [Background] Kennedy EP, Rosato EL, Sauter PK, Rosenberg LM, Doria C, Marino IR, Chojnacki KA, Berger AC, Yeo CJ. Initiation of a critical pathway for pancreaticoduodenectomy at an academic institution--the first step in multidisciplinary team building. J Am Coll Surg. 2007 May;204(5):917-23; discussion 923-4. doi: 10.1016/j.jamcollsurg.2007.01.057. PMID 17481510
- [Background] Lassen K, Coolsen MM, Slim K, Carli F, de Aguilar-Nascimento JE, Schafer M, Parks RW, Fearon KC, Lobo DN, Demartines N, Braga M, Ljungqvist O, Dejong CH; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care for pancreaticoduodenectomy: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. World J Surg. 2013 Feb;37(2):240-58. doi: 10.1007/s00268-012-1771-1. No abstract available. PMID 22956014
- [Background] Lassen K, Soop M, Nygren J, Cox PB, Hendry PO, Spies C, von Meyenfeldt MF, Fearon KC, Revhaug A, Norderval S, Ljungqvist O, Lobo DN, Dejong CH; Enhanced Recovery After Surgery (ERAS) Group. Consensus review of optimal perioperative care in colorectal surgery: Enhanced Recovery After Surgery (ERAS) Group recommendations. Arch Surg. 2009 Oct;144(10):961-9. doi: 10.1001/archsurg.2009.170. PMID 19841366
- [Background] Stergiopoulou A, Birbas K, Katostaras T, Mantas J. The effect of interactive multimedia on preoperative knowledge and postoperative recovery of patients undergoing laparoscopic cholecystectomy. Methods Inf Med. 2007;46(4):406-9. doi: 10.1160/me0406. PMID 17694232
- [Background] Varadhan KK, Neal KR, Dejong CH, Fearon KC, Ljungqvist O, Lobo DN. The enhanced recovery after surgery (ERAS) pathway for patients undergoing major elective open colorectal surgery: a meta-analysis of randomized controlled trials. Clin Nutr. 2010 Aug;29(4):434-40. doi: 10.1016/j.clnu.2010.01.004. Epub 2010 Jan 29. PMID 20116145